CLINICAL TRIAL: NCT02168140
Title: Phase I Dose-Escalation Study of CPI-613, in Combination With Bendamustine, in Patients With Relapsed or Refractory T-Cell Non-Hodgkin Lymphoma or Classic Hodgkin Lymphoma
Brief Title: CPI-613 and Bendamustine Hydrochloride in Treating Patients With Relapsed or Refractory T-Cell Non-Hodgkin Lymphoma or Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00028206; NCI-2014-01281 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 28314 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2023-12

CONDITIONS: Adult Lymphocyte Depletion Hodgkin Lymphoma; Adult Lymphocyte Predominant Hodgkin Lymphoma; Adult Mixed Cellularity Hodgkin Lymphoma; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Adult Nodular Sclerosis Hodgkin Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Hepatosplenic T-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; T-cell Adult Acute Lymphoblastic Leukemia; T-cell Large Granular Lymphocyte Leukemia
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Leukemia, Large Granular Lymphocytic | interventions — devimistat; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CPI-613 and bendamustine hydrochloride) (Experimental): Patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-4 of week 1 and on days 1 and 4 of weeks 2 and 3. Patients also receive bendamustine hydrochloride IV over 30 minutes on days 4 and 5 of week 1. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 6,8-bis(benzylthio)octanoic acid; Drug: bendamustine hydrochloride

INTERVENTIONS:
Drug: 6,8-bis(benzylthio)octanoic acid — Given IV
  Other Names: alpha-lipoic acid analogue CPI-613; CPI-613
Drug: bendamustine hydrochloride — Given IV
  Other Names: bendamustin hydrochloride; bendamustine; cytostasan hydrochloride; Treanda

SUMMARY:
This phase I trial studies the side effects and best dose of CPI-613 when given together with bendamustine hydrochloride in treating patients with relapsed or refractory T-cell non-Hodgkin lymphoma or Hodgkin lymphoma. CPI-613 may kill cancer cells by turning off their mitochondria, which are used by cancer cells to produce energy and are the building blocks needed to make more cancer cells. By shutting off mitochondria, CPI-613 may deprive the cancer cells of energy and other supplies needed to survive and grow. Drugs used in chemotherapy, such as bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving CPI-613 with bendamustine hydrochloride may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of CPI-613 [6,8-bis(benzylthio)octanoic acid], when used in combination with bendamustine (bendamustine hydrochloride) in patients with relapsed and refractory classic Hodgkin lymphoma (HL) or T-cell non-Hodgkin lymphoma (NHL) who have or have not received hematopoietic cell transplant.

SECONDARY OBJECTIVES:

I. To evaluate response rate (RR) and disease control rate (DCR), derived from the modified International Work Group (IWG) criteria and International Cutaneous Lymphoma (Olsen criteria) for cutaneous lymphomas.

II. To evaluate overall survival (OS) and progression-free survival (PFS), and possible correlation between RR and DCR derived from modified IWF criteria vs. OS and PFS.

III. To evaluate assessment of bone marrow biopsy, and possible correlation between complete response (CR) vs. bone marrow biopsy assessment (e.g., clear of infiltration of leukemic cells according to morphology, and/or negative on leukemic cells according to immunohistochemistry).

IV. To evaluate safety of CPI-613 + bendamustine combination.

OUTLINE: This is a dose-escalation study of 6,8-bis(benzylthio)octanoic acid.

Patients receive 6,8-bis(benzylthio)octanoic acid intravenously (IV) over 2 hours on days 1-4 of week 1 and on days 1 and 4 of weeks 2 and 3. Patients also receive bendamustine hydrochloride IV over 30 minutes on days 4 and 5 of week 1. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed T-cell NHL or classic HL (i.e., nodular sclerosis HL, mixed cellularity HL, lymphocyte rich classic HL, and lymphocyte depleted HL) that has relapsed from, or is refractory to, all standard therapies (including autologous transplantation) known to provide clinical benefit, but have not been treated with bendamustine for their lymphoma
* Must have measurable disease (e.g., a tumor mass > 1 cm)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Expected survival > 3 months
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists
* At least 2 weeks must have elapsed from any prior surgery
* Aspartate aminotransferase (AST/serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x upper normal limit (UNL), alanine aminotransferase (ALT/serum glutamate pyruvate transaminase [SGPT]) =< 3 x UNL (=< 5 x UNL if liver metastases present)
* Bilirubin =< 1.5 x UNL
* Serum creatinine =< 1.5 mg/dL or 133 µmol/L
* "International normalized ratio" or INR must be =< 1.5
* No evidence of active infection and no serious infection within the past month
* Mentally competent, ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

* Known cerebral metastases, central nervous system (CNS) or epidural tumor
* Having "currently active" second malignancy unrelated to HL or NHL, unless they have completed anti-cancer therapy, are in complete response and are considered by their physicians to be at less than 30% risk of relapse
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication, within the past 2 weeks prior to initiation of treatment with study drugs
* Serious medical illness that would potentially increase patients' risk for toxicity
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease)
* History of abdominal fistula or gastrointestinal perforation =< 6 months prior to treatment with study drugs
* Pregnant women, or women of child-bearing potential not using reliable means of contraception
* Lactating females
* Fertile men unwilling to practice contraceptive methods during the study period
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
* Unwilling or unable to follow protocol requirements
* Active heart disease including but not limited to symptomatic congestive heart failure, symptomatic coronary artery disease, symptomatic angina pectoris, symptomatic myocardial infarction or symptomatic congestive heart failure
* Patients with a history of myocardial infarction that is < 3 months prior to registration
* Evidence of active infection, or serious infection within the past month
* Patients with known human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Patients who have received cancer immunotherapy of any type within the past 2 weeks prior to initiation of CPI-613 treatment
* Requirement for immediate palliative treatment of any kind including surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
MTD of 6,8-bis(benzylthio)octanoic acid when used in combination with bendamustine hydrochloride, defined as the dose level immediately below the dose level that induced a dose-limiting toxicity in < 2 patients | Up to 28 days
  Graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.

OTHER OUTCOMES:
RR, derived from the modified IWG criteria and the International Cutaneous Lymphoma (Olsen criteria) for cutaneous lymphoma | Up to 3 years
  RR and its 95% confidence interval will be assessed. RR and the possible correlation between RR and DCR vs. OS and PFS will be evaluated.
DCR, derived from the modified IWG criteria and the International Cutaneous Lymphoma (Olsen criteria) for cutaneous lymphoma | Up to 3 years
  DCR and its 95% confidence interval will be assessed. DCR and the possible correlation between RR and DCR vs. OS and PFS will be evaluated.
OS | Time from first dose of 6,8-bis(benzylthio)octanoic acid to death by any cause, assessed up to 3 years
  OS curves will be plotted using Kaplan-Meier methods. OS and the possible correlation between RR and DCR vs. OS and PFS will be evaluated.
PFS | Time from first dose of 6,8-bis(benzylthio)octanoic acid to disease progression, assessed up to 3 years
  PFS curves will be plotted using Kaplan-Meier methods and median PFS will be examined. PFS and the possible correlation between RR and DCR vs. OS and PFS will be evaluated.
Bone marrow biopsy assessment | After course 6 (168 days)
  Bone marrow and possible correlation between CR vs. bone marrow biopsy assessments such as clear of infiltration of leukemic cells according to morphology, and/or negative on leukemic cells according to immunohistochemistry will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Rakhee Vaidya, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina
  - Abramson Cancer Center, Philadelphia, Pennsylvania

DOCUMENTS (1):
  • Informed Consent Form (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT02168140/ICF_000.pdf